CLINICAL TRIAL: NCT01238380
Title: Using Pharmacogenetics to Improve Treatment in Early-onset Diabetes
Acronym: UNITED
Status: Completed | Type: Observational
Sponsor: University of Exeter (Other)
Collaborators: University of Dundee (Other); Wellcome Trust (Other); Department of Health, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: REC 10/H0106/63; HICF-1009-041 (Other Grant/Funding Number: Wellcome Trust and Department of Health)
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Diabetes
Keywords: Monogenic diabetes; HNF1A; HNF4A; GCK; genetic testing; health economic model
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples with DNA and plasma samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diabetes diagnosed under 30 years: Patients currently under 50 years of age diagnosed with diabetes under 30 years.
  Interventions: Other: patient care pathway

INTERVENTIONS:
Other: patient care pathway — Stage 1: Urinary c-peptide creatinine ratio (UCPCR); if positive progress to Stage 2.
  Stage 2: Pancreatic auto-antibodies measurement (GAD65 & IA2); if negative progress to genetic testing.
  Genetic testing for HNF1A, HNF4A, GCK. If positive, progress to Stage 3.
  Stage 3: review and potential change of diabetes treatment. Monitor success via use of three standardised health and quality of life questionnaires and Hba1c pre-treatment change and at 1, 3, 6 and 12 months post-treatment change.

SUMMARY:
Monogenic diabetes is an unusual form of diabetes. It usually presents in patients under the age of 30, so is often misdiagnosed as Type 1 diabetes which is more common. Patients with monogenic diabetes can often be treated with tablets rather than insulin injections, leading to better control of their diabetes, and fewer side-effects and complications. Less than 5% of people with monogenic diabetes in the UK have been identified, meaning up to 20,000 patients may still be misdiagnosed and receiving inappropriate treatment. We want to identify the best way of ensuring that people diagnosed with diabetes under the age of 30 have all the necessary tests to ensure they have the correct treatment for their particular type of diabetes. A small number of people may, as part of this study, be found to have a specific genetic cause of their diabetes and in these cases we will measure the success and benefits of changing their treatment, usually from insulin injections to sulphonylurea tablets.

DETAILED DESCRIPTION:
Aim:The aim of this project is to identify a patient pathway which ensures that patients with young-onset diabetes (diagnosed <30 years) have a systematic series of investigations which allow for appropriate genetic testing and hence appropriate alteration of therapy if required.

Objectives:

1. To establish and test a care pathway to detect monogenic diabetes in patients with diabetes diagnosed before the age of 30 years and currently under the age of 50 years. This will indicate the prevalence of monogenic diabetes.
2. To measure the success, cost and potential economic benefit of changing the treatment of those patients identified with monogenic diabetes from their initial therapy, typically insulin injections, to appropriate treatment, usually oral sulphonylureas.
3. To obtain the necessary data to enable the development of an appropriate health economic model.

This project will provide evidence for a cost-based model for a systematic care pathway for the diagnosis and treatment of diabetes diagnosed < 30 years. The pathway will select subjects by clinical, biochemical (urinary C peptide) and immunological (pancreatic autoantibodies) criteria for genetic testing. The present approach relies on clinicians recognising the possibility of a monogenic cause and arranging genetic testing. In the UK less than 5% of the estimated cases of monogenic diabetes have been identified and this means that up to 20,000 diabetic patients are receiving inappropriate treatment. Patients confirmed by molecular genetic testing to have monogenic diabetes may benefit from changing from insulin and other therapies, to treatment with sulphonylurea tablets or diet alone. Systematic targeted use of molecular genetic testing in young-onset diabetes will result in stratified treatment according to aetiology with improved efficacy, quality of life and long term complication risk, while reducing side effects and cost.

This project aims to develop a pathway of testing in patients diagnosed under the age of 30 years, to identify those who should receive genetic testing. This will consist of three stages: 1) a urine test that can determine if a patient is making their own insulin; 2) for those who are making their own insulin, a further blood test will be carried out testing for antibodies which are seen in Type 1 diabetes; 3) in those who are negative for the antibodies, a genetic test will be carried out to determine whether they have monogenic diabetes. Individuals who are found to have monogenic diabetes may have their treatment changed.

Project Plan This project will be based in Exeter and undertaken in collaboration with colleagues at Ninewells Hospital Trust and the University of Dundee in Scotland. Within the defined geographical regions of Tayside and Devon, all patients with diabetes diagnosed under 30 years of age, and who are currently aged less than 50 years, will be invited to participate in the study. We estimate that from a total population of 800,000 (400,000 in Devon and 400,000 in Tayside) a potential group of 3,000 patients will be identified, of which approximately 90% (n=2700) are likely to be insulin treated.

Initial procedure following recruitment:

Participants will be provided with a written patient information sheet, a consent form, a urine sample container and written instructions for sample collection. Baseline data will be collected either face to face or by telephone by a member of the research team. Participants will be asked to provide a single urine sample 2 hours after their main meal of the day. Baseline data on all subjects will include age, age at diagnosis, duration of diabetes, height, weight, initial/current treatment, and any family history of diabetes. Permission to access their medical records will be obtained in order to clarify or confirm relevant clinical data. The participant will be asked to return the completed consent form and the urine sample to the research team or through routine NHS courier service if samples are returned to local GPs.

In Tayside, patients with a clinical diagnosis of Type 1 diabetes, aged over 16 years old, will initially be recruited into the Scottish Diabetes Research Network Type 1 Diabetes Bioresource (Ethics ref: 10/S140243). Those diagnosed under 30 years of age, who are currently aged less than 50 years old, will be asked to return a post-meal urine sample to the research team and will proceed as for other UNITED study participants.

Following this initial urine test, participants found to be UCPCR negative will be informed of their result via a standardised letter. This will complete their involvement with the project.

Participants found to be UCPCR positive will be informed of their result by a member of the research team and given the opportunity to discuss the implications for the next stage of the project.

1. UCPCR positive patients:

   Participants will be invited to the Peninsula Clinical Research Facility (PCRF), Ninewells Clinical Research Centre (NCRC), or a suitable local venue where blood samples for pancreatic auto-antibodies (GAD and IA2), DNA extraction and HbA1c will be taken by a member of the research team.

   Following this initial antibody screen those participants found to be antibody positive will be informed of their result via a standardised letter (Stage2/GADpos/Vs1/0810). This will complete their involvement with the project.

   Those participants found to be antibody negative will be informed of their result in person by a member of the research team and given the opportunity to discuss the implications for the next stage of the project.
2. UCPCR positive and Antibody negative patients:

   Participants who are now known to be UCPCR positive and antibody negative will be offered genetic screening for monogenic diabetes. Information will be provided by the research team, who will be trained in genetic counselling, about the implications of genetic testing and the possible consequences of a positive or negative result for the individual and in the case of a positive result the implications for other family members.

   Those participants found to be negative following genetic screening will be informed of their result by a member of the research team. This will be followed up by a standardised letter (Stage2/neg-gen-test/Vs1/0810) and this will complete their involvement with the project.

   Those participants with a positive result following genetic screening will be informed of their results in person by a member of the research team, and given the opportunity to discuss the implications for the next stage of the project.
3. The participants in the subsequent stages of the project are those now defined as:

   * UCPCR positive
   * antibody negative
   * confirmed to have a diagnosis of monogenic diabetes following molecular genetic testing.

It is anticipated that participants may require a review and revision of their current treatment. This review will be by the NHS Clinician who manages the participant's diabetes. They will be informed by NHS Clinical experts in monogenic diabetes.

Transfer of patients identified with monogenic diabetes to alternative treatment Following the review, all participants who are not on the appropriate treatment will be transferred to sulphonylureas for HNF1A/HNF4A and no treatment for GCK mutations. As these subjects will only be identified after they have gone through the screening program, in order to increase numbers in this part of the project and to enable accurate assessment of potential costs and benefits of the transfer, we will also recruit patients for this assessment by including patients with monogenic diabetes diagnosed outside of the project. At present the diagnostic lab is identifying approximately 10 new UK patients per month. Referring Clinicians will be sent written information on the project via a standardised letter (MODY referring Clinician covering letter - Vs1/0810) which will accompany test result. Participants identified through this route will allow us to recruit additional patients to ensure that there are sufficient data to achieve good confidence limits for the estimates required for the future development of a health economic model.

The assessment of success of treatment transfer on glycaemic control and quality of life:

Participants will be asked to fill in baseline standardised questionnaires (ADDQoL, EQ5D and the DTSQs) to assess patient reported outcomes including: the impact of diabetes on their quality of life, their current health status and their treatment satisfaction while on their current treatment. Child participants be asked to fill in age appropriate versions of the study questionnaires: the ADDQoL-Teen,(for teenagers up to 16 years), the ADDQoL-Junior (for 5-8 year olds), ADDQoL- Junior Plus (for 9-12 year olds), the EQ-5D youth/children (age 7-12 years), DTSQ-Teen (teenagers up to 16 years of age). Where appropriate those with parental responsibility will be asked to provide information by completing the DTSQ-Parent.

Following treatment change, participants will be followed up by the diabetes specialist research nurses as often as the participant requires in order to assess their treatment needs, or to provide emotional support. This may initially be daily for the first week, then tailing off gradually as the individual becomes confident on their new treatment and their blood glucose levels stablise. The timings will be dependent on individual need.

Post treatment questionnaire follow up:

1 month - repeat DTSQs and EQ5D 6 month - repeat DTSQs and EQ5D and ADDQoL 12 months repeat DTSQs followed by DTSQc, EQ5D and ADDQoL.

Blood samples for HbA1C will be taken at 3, 6 and 12 months.

Participant involvement in the study will be complete 12 months following initial treatment change. During this 12 month period the clinical care of these participants will remain the responsibility of their NHS clinician. These clinicians will be informed by NHS experts in monogenic diabetes.

Development of Heath Economic model prototype A health economic model will be developed to compare the likely costs and effects of the new care pathway with current practice. This will be informed by a systematic review of the current relevant economic literature and build on existing economic models for diabetes. It will also be informed by results from this project.

Funding:This study has been funded by a grant from the Health Innovation Challenge Fund (HICF) which is a joint venture between the Department of Health and the Wellcome Trust. Project funding will be administered by the University of Exeter. A collaboration agreement between the University of Exeter and the University of Dundee will be established to determine the distribution of funding between the two organisations.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of diabetes
* diagnosed under 30 years of ages
* current age less than 50 years
* willing and able to provide informed consent.

Exclusion Criteria:

* age over 50 years
* age at diagnosis over 30 years
* adult with incapacity to consent
* child with incapacity to assent

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients currently under the age of 50 years, diagnosed under the age of 30years, from South-West England and Tayside, Scotland, UK.
Sampling Method: Non-Probability Sample
Enrollment: 1916 (Actual)
Dates: Start 2010-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Identification of patients with monogenic diabetes | Within 4 years from start of project
  The aim of this project is to identify the prevalence of patients with monogenic diabetes resulting from mutations in the HNF1A/HNF4A/GCK genes, amongst patients with early-onset diabetes, diagnosed less than 30 years.

SECONDARY OUTCOMES:
To examine the impact of making a diagnosis of monogenic diabetes on patients' treatment, glucose control and quality of life. | Within 4 years of the project start date.
  To measure the impact of making a molecular genetic diagnosis of monogenic diabetes by examining at baseline, 1 month, 6 months and 12 months the following parameters:
  i) treatment - both type and dose; ii) glucose control - measured by HbA1c at 3, 6 and 12 months post-treatment change; iii) quality of life - by appropriate protocols.
To develop a health economic model of the care pathway leading to testing of monogenic diabetes. | Within 4 years of the project start date.
  To develop a health economic model that can measure the success, cost and potential economic benefit of using the care pathway to identify patients with monogenic diabetes and potentially change their treatment. This will allow assessment of when testing is appropriate on health economic grounds.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T Hattersley, Principal Investigator — Peninsula NIHR Clinical Research Facility, Peninsula Medical School, University of Exeter, Barrack Rd, Exeter, EX2 5DW
Locations (3):
- United Kingdom (3):
  - Peninsula NIHR Clinical Research Facility, Peninsula Medical School, Barrack Rd,, Exeter, Devon
  - Peninsula College of Medicine & Dentistry, University of Plymouth, John Bull Building, Tamar Science Park,, Plymouth, Devon
  - Biomedical Research Institute, University of Dundee,, Dundee

REFERENCES:
- [Background] Shields BM, Hicks S, Shepherd MH, Colclough K, Hattersley AT, Ellard S. Maturity-onset diabetes of the young (MODY): how many cases are we missing? Diabetologia. 2010 Dec;53(12):2504-8. doi: 10.1007/s00125-010-1799-4. Epub 2010 May 25. PMID 20499044
- [Background] McDonald TJ, Knight BA, Shields BM, Bowman P, Salzmann MB, Hattersley AT. Stability and reproducibility of a single-sample urinary C-peptide/creatinine ratio and its correlation with 24-h urinary C-peptide. Clin Chem. 2009 Nov;55(11):2035-9. doi: 10.1373/clinchem.2009.129312. Epub 2009 Aug 27. PMID 19713273
- [Background] Shepherd M, Shields B, Ellard S, Rubio-Cabezas O, Hattersley AT. A genetic diagnosis of HNF1A diabetes alters treatment and improves glycaemic control in the majority of insulin-treated patients. Diabet Med. 2009 Apr;26(4):437-41. doi: 10.1111/j.1464-5491.2009.02690.x. PMID 19388975
- [Background] Ellard S, Bellanne-Chantelot C, Hattersley AT; European Molecular Genetics Quality Network (EMQN) MODY group. Best practice guidelines for the molecular genetic diagnosis of maturity-onset diabetes of the young. Diabetologia. 2008 Apr;51(4):546-53. doi: 10.1007/s00125-008-0942-y. Epub 2008 Feb 23. PMID 18297260
- [Background] Pearson ER, Pruhova S, Tack CJ, Johansen A, Castleden HA, Lumb PJ, Wierzbicki AS, Clark PM, Lebl J, Pedersen O, Ellard S, Hansen T, Hattersley AT. Molecular genetics and phenotypic characteristics of MODY caused by hepatocyte nuclear factor 4alpha mutations in a large European collection. Diabetologia. 2005 May;48(5):878-85. doi: 10.1007/s00125-005-1738-y. Epub 2005 Apr 14. PMID 15830177
- [Background] Pearson ER, Starkey BJ, Powell RJ, Gribble FM, Clark PM, Hattersley AT. Genetic cause of hyperglycaemia and response to treatment in diabetes. Lancet. 2003 Oct 18;362(9392):1275-81. doi: 10.1016/S0140-6736(03)14571-0. PMID 14575972
- [Derived] Grace SL, Cooper A, Jones AG, McDonald TJ. Zinc transporter 8 autoantibody testing requires age-related cut-offs. BMJ Open Diabetes Res Care. 2021 Aug;9(1):e002296. doi: 10.1136/bmjdrc-2021-002296. PMID 34348918
- [Derived] Peters JL, Anderson R, Shields B, King S, Hudson M, Shepherd M, McDonald TJ, Pearson E, Hattersley A, Hyde C. Strategies to identify individuals with monogenic diabetes: results of an economic evaluation. BMJ Open. 2020 Mar 18;10(3):e034716. doi: 10.1136/bmjopen-2019-034716. PMID 32193268
- [Derived] Shields BM, Shepherd M, Hudson M, McDonald TJ, Colclough K, Peters J, Knight B, Hyde C, Ellard S, Pearson ER, Hattersley AT; UNITED study team. Population-Based Assessment of a Biomarker-Based Screening Pathway to Aid Diagnosis of Monogenic Diabetes in Young-Onset Patients. Diabetes Care. 2017 Aug;40(8):1017-1025. doi: 10.2337/dc17-0224. PMID 28701371
- See also: website providing information regarding monogenic diabetes — http://www.diabetesgenes.org